CLINICAL TRIAL: NCT00853047
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Ascending, Multidose Study To Determine Safety and Tolerability of Orally Administered LX1606 in Subjects With Symptomatic Carcinoid Syndrome Refractory to Stable-Dose Octreotide Long-Acting Release Depot Therapy
Brief Title: Study of Telotristat Etiprate (LX1606) in Participants With Symptomatic Carcinoid Syndrome Not Managed by Stable-Dose Octreotide Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LX1606.1-202-CS; LX1606.202 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2009-02-25; First posted 2009-02-27 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-10

CONDITIONS: Carcinoid Syndrome
MeSH Terms: conditions — Serotonin Syndrome | interventions — telotristat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Telotristat Etiprate 150 mg Core Phase (Experimental): Telotristat etiprate capsules,150 mg orally 3 times daily for 28 days in the double-blind treatment period (core phase) in combination with stable-dose octreotide long-acting release (LAR) depot therapy given once per month. Upon completion of 28-days of treatment, participants were eligible to enter the optional open-label extension period.
  Interventions: Drug: Telotristat etiprate; Drug: Octreotide LAR Depot
- Telotristat Etiprate 250 mg Core Phase (Experimental): Telotristat etiprate capsules, 250 mg orally 3 times daily for 28 days in the double-blind treatment period in combination with stable-dose octreotide LAR depot therapy given once per month. Upon completion of 28-days of treatment, participants were eligible to enter the optional open-label extension period.
  Interventions: Drug: Telotristat etiprate; Drug: Octreotide LAR Depot
- Telotristat Etiprate 350 mg Core Phase (Experimental): Telotristat etiprate capsules, 350 mg orally 3 times daily for 28 days in the double-blind treatment period in combination with stable-dose octreotide LAR depot therapy given once per month. Upon completion of 28-days of treatment, participants were eligible to enter the optional open-label extension period.
  Interventions: Drug: Telotristat etiprate; Drug: Octreotide LAR Depot
- Telotristat Etiprate 500 mg Core Phase (Experimental): Telotristat etiprate capsules, 500 mg orally 3 times daily for 28 days in the double-blind treatment period in combination with a stable-dose octreotide LAR depot therapy given once per month. Upon completion of 28-days of treatment, participants were eligible to enter the optional open-label extension period.
  Interventions: Drug: Telotristat etiprate; Drug: Octreotide LAR Depot
- Placebo Core Phase (Experimental): Placebo-matching telotristat etiprate capsules, orally 3 times daily for 28 days in the double-blind treatment period in combination with stable-dose octreotide LAR depot therapy given once per month. Upon completion of 28-days of treatment, participants were eligible to receive telotristat etiprate in the optional open-label extension period.
  Interventions: Drug: Octreotide LAR Depot; Drug: Placebo
- Telotristat Etiprate Open-Label Extension Phase (Experimental): Telotristat etiprate at assigned dose level for 8 weeks in combination with stable-dose octreotide LAR depot therapy given once per month in the open-label extension period. Upon completion of the 8-week period, participants could enter an additional extension period of 172 weeks, receiving telotristat etiprate at the assigned dose or maximum tolerated dose (500 mg 3 times daily).
  Interventions: Drug: Telotristat etiprate; Drug: Octreotide LAR Depot

INTERVENTIONS:
Drug: Telotristat etiprate — Telotristat etiprate capsules; orally 3 times daily.
  Other Names: LX1606
  Arms: Telotristat Etiprate 150 mg Core Phase; Telotristat Etiprate 250 mg Core Phase; Telotristat Etiprate 350 mg Core Phase; Telotristat Etiprate 500 mg Core Phase; Telotristat Etiprate Open-Label Extension Phase
Drug: Octreotide LAR Depot — A stable-dose octreotide LAR depot therapy; administered subcutaneously once per month.
Drug: Placebo — Placebo-matching telotristat etiprate capsules; orally 3 times daily.
  Arms: Placebo Core Phase

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of telotristat etiprate (LX1606) versus a placebo control in participants with symptomatic carcinoid syndrome not managed by stable-dose long-acting octreotide therapy. Following determination of the maximally tolerated or effective dose, cohort expansion will occur to confirm effect on symptoms and safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, aged 18 and older
* Biopsy-proven metastatic carcinoid tumor of the gastrointestinal (GI) tract with disease extent confirmed by computed tomography (CT), magnetic resonance imaging (MRI), or radionuclide imaging
* Symptoms not managed by stable-dose long-acting octreotide therapy (≥4 bowel movements per day)
* Ability to provide written informed consent

Exclusion Criteria:

* ≥12 high volume, watery bowel movements per day associated with a clinical syndrome of volume contraction, dehydration, or hypotension compatible with a "pancreatic cholera"-type clinical syndrome
* Sponsor-unacceptable clinical laboratory values for hematology and liver function tests at screening
* Karnofsky status ≤70% - unable to care for self
* Surgery within 60 days prior to screening
* A history of short bowel syndrome
* Life expectancy <12 months
* History of substance or alcohol abuse within 2 years prior to screening
* Previous exposure to a tryptophan hydroxylase (TPH) inhibitor
* Administration of any investigational drug within 30 days of screening or any therapeutic protein or antibody within 90 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Lapuerta, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (9):
- United States (9):
  - Hematology Oncology Services of Arkansas, Little Rock, Arkansas
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - St. Francis Medical Group Oncology and Hematology Specialists, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - UT M.D. Anderson Cancer Center, Houston, Texas
  - Texas Oncology - McAllen, McAllen, Texas
  - Texas Oncology - Weslaco, Weslaco, Texas

REFERENCES:
- [Derived] Gelhorn HL, Kulke MH, O'Dorisio T, Yang QM, Jackson J, Jackson S, Boehm KA, Law L, Kostelec J, Auguste P, Lapuerta P. Patient-reported Symptom Experiences in Patients With Carcinoid Syndrome After Participation in a Study of Telotristat Etiprate: A Qualitative Interview Approach. Clin Ther. 2016 Apr;38(4):759-68. doi: 10.1016/j.clinthera.2016.03.002. Epub 2016 Mar 31. PMID 27041406
- [Derived] Kulke MH, O'Dorisio T, Phan A, Bergsland E, Law L, Banks P, Freiman J, Frazier K, Jackson J, Yao JC, Kvols L, Lapuerta P, Zambrowicz B, Fleming D, Sands A. Telotristat etiprate, a novel serotonin synthesis inhibitor, in patients with carcinoid syndrome and diarrhea not adequately controlled by octreotide. Endocr Relat Cancer. 2014 Oct;21(5):705-14. doi: 10.1530/ERC-14-0173. Epub 2014 Jul 10. PMID 25012985

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 23 participants were enrolled in the Core Phase (ie, Screening and Double-blind Treatment Period) from 11 sites, including 1 satellite site, in the United States. 19 participants entered the Open-label Extension Phase.
Groups:
- Placebo Core Phase: Participants received placebo-matching telotristat etiprate capsules, orally 3 times daily for 28 days in the double-blind treatment period (core phase) in combination with stable-dose octreotide long-acting release (LAR) depot therapy given once per month. Upon completion of 28-days of treatment, participants were eligible to receive telotristat etiprate in the optional open-label extension period.
- Telotristat Etiprate 150 mg Core Phase: Participants received telotristat etiprate capsules,150 mg orally 3 times daily for 28 days in the double-blind treatment period in combination with stable-dose octreotide LAR depot therapy given once per month. Upon completion of 28-days of treatment, participants were eligible to enter the optional open-label extension period.
- Telotristat Etiprate 250 mg Core Phase: Participants received telotristat etiprate capsules, 250 mg orally 3 times daily for 28 days in the double-blind treatment period in combination with stable-dose octreotide LAR depot therapy given once per month. Upon completion of 28-days of treatment, participants were eligible to enter the optional open-label extension period.
- Telotristat Etiprate 350 mg Core Phase: Participants received telotristat etiprate capsules, 350 mg orally 3 times daily for 28 days in the double-blind treatment period in combination with stable-dose octreotide LAR depot therapy given once per month. Upon completion of 28-days of treatment, participants were eligible to enter the optional open-label extension period.
- Telotristat Etiprate 500 mg Core Phase: Participants received telotristat etiprate capsules, 500 mg orally 3 times daily for 28 days in the double-blind treatment period in combination with a stable-dose octreotide LAR depot therapy given once per month. Upon completion of 28-days of treatment, participants were eligible to enter the optional open-label extension period.
- Telotristat Etiprate Open-Label Extension Phase: Participants received telotristat etiprate at assigned dose level for 8 weeks in combination with stable-dose octreotide LAR depot therapy given once per month in the open-label extension period. Upon completion of the 8-week period, participants could enter an additional extension period of 172 weeks, receiving telotristat etiprate at the assigned dose or maximum tolerated dose (500 mg 3 times daily).
Period: Core Phase
Arm/Group | Placebo Core Phase | Telotristat Etiprate 150 mg Core Phase | Telotristat Etiprate 250 mg Core Phase | Telotristat Etiprate 350 mg Core Phase | Telotristat Etiprate 500 mg Core Phase | Telotristat Etiprate Open-Label Extension Phase
Started | 5 | 3 | 3 | 3 | 9 | 0
Completed | 5 | 3 | 3 | 2 | 9 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant Request | 0 | 0 | 0 | 1 | 0 | 0
Period: Open-Label Extension Phase
Arm/Group | Placebo Core Phase | Telotristat Etiprate 150 mg Core Phase | Telotristat Etiprate 250 mg Core Phase | Telotristat Etiprate 350 mg Core Phase | Telotristat Etiprate 500 mg Core Phase | Telotristat Etiprate Open-Label Extension Phase
Started | 0 | 0 | 0 | 0 | 0 | 19 (19 of the 22 participants who completed the Core Phase entered the optional Open-Label Extension.)
Completed 8-week Extension Period | 0 | 0 | 0 | 0 | 0 | 16
Completed | 0 | 0 | 0 | 0 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 17
Not completed — Participant Request | 0 | 0 | 0 | 0 | 0 | 7
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Transfer to LX1606-302 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Investigator Decision | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Population: The Safety Set, Core Phase included all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Core Phase | Telotristat Etiprate 150 mg Core Phase | Telotristat Etiprate 250 mg Core Phase | Telotristat Etiprate 350 mg Core Phase | Telotristat Etiprate 500 mg Core Phase | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 9 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (11.72) | 51.7 (8.08) | 61.0 (16.09) | 52.7 (9.81) | 65.7 (9.94) | 60.8 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 2 | 4 | 12
  Male | 3 | 0 | 2 | 1 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 1
  White | 5 | 2 | 3 | 3 | 9 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE) and Any Drug-related TEAE in the Core Phase
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. A TEAE was an AE reported after the first dose of randomized treatment on Day 1.
Time Frame: Up to 4 Weeks Core Phase
Population: The Safety Set Core Phase included all participants who received at least one dose of study drug in the core phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Core Phase | Telotristat Etiprate 150 mg Core Phase | Telotristat Etiprate 250 mg Core Phase | Telotristat Etiprate 350 mg Core Phase | Telotristat Etiprate 500 mg Core Phase
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 9
Participants
  Any TEAE | 4 | 3 | 3 | 2 | 9
  Related TEAEs | 3 | 3 | 0 | 2 | 6

2. Primary Outcome: Number of Participants With Any TEAE in the Open-Label Extension Phase
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A TEAE was an AE reported after receiving treatment.
Time Frame: Up to 180 weeks in the open-label extension phase
Population: The Safety Set Extension Period included all participants who received at least one dose of study drug in the open-label extensions phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Telotristat Etiprate Open-Label Extension Phase
Number analyzed (Participants) | 19
Participants | 18

3. Secondary Outcome: Change From Baseline in Mean Number of Bowel Movements (BMs) Per Day
Description: Participants recorded the number of BMs per day in a daily diary. The total number of BMs per day were averaged over the 4-week period. A negative change from Baseline indicates improvement.
Time Frame: Baseline to Week 4
Population: Participants from the modified Intent to Treat (mITT) Set, Core Phase, all participants who received any fraction of a dose of study drug and had at least 1 week of data recorded in the daily diary after receiving study drug, with data available for analysis.
Measure: Mean (Standard Deviation); unit: bowel movements/day
Arm/Group | Placebo Core Phase | Telotristat Etiprate 150 mg Core Phase | Telotristat Etiprate 250 mg Core Phase | Telotristat Etiprate 350 mg Core Phase | Telotristat Etiprate 500 mg Core Phase
Number analyzed (Participants) | 4 | 3 | 3 | 1 | 7
bowel movements/day | 0.82 (0.435) | -1.37 (1.514) | -2.17 (2.259) | -0.20 (0) | -0.71 (2.048)

4. Secondary Outcome: Change From Baseline in Weekly Mean Stool Form
Description: Participants recorded stool form in a daily diary using a 6-point scale (0-none,1-hard, 2-firm, 3-soft, 4-loose, 5-watery). A negative change from Baseline indicates improvement.
Time Frame: Baseline to Week 4
Population: Participants from the mITT Set Core Phase, all participants who received any fraction of a dose of study drug and had at least 1 week of data recorded in the daily diary after receiving study drug, with data available for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Core Phase | Telotristat Etiprate 150 mg Core Phase | Telotristat Etiprate 250 mg Core Phase | Telotristat Etiprate 350 mg Core Phase | Telotristat Etiprate 500 mg Core Phase
Number analyzed (Participants) | 4 | 3 | 2 | 1 | 7
units on a scale | -0.07 (0.222) | -0.50 (0.755) | 0.00 (0.141) | 0.00 (0) | -0.17 (0.579)

5. Secondary Outcome: Change From Baseline in Percentage of Days Per Week Experiencing a Sensation of Urgency to Defecate
Description: Participants recorded the sensation of urgency to defecate (Yes or No) in a daily diary. A negative change from Baseline indicates improvement.
Time Frame: Baseline to Week 4
Population: Participants from the mITT Set Core Phase, all participants who received any fraction of a dose of study drug and had at least 1 week of data recorded in the daily diary after receiving study drug with data available for analysis.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo Core Phase | Telotristat Etiprate 150 mg Core Phase | Telotristat Etiprate 250 mg Core Phase | Telotristat Etiprate 350 mg Core Phase | Telotristat Etiprate 500 mg Core Phase
Number analyzed (Participants) | 4 | 3 | 3 | 1 | 7
percentage of days | -2.72 (5.164) | -34.43 (47.261) | -32.13 (28.328) | 0.00 (0) | -8.49 (15.742)

6. Secondary Outcome: Change From Baseline in Number of Cutaneous Flushing Episodes
Description: Participants recorded the number of daily flushing episodes per day in a daily diary. The total number of flushing episodes per day were averaged over the 4-week period. A negative change from Baseline indicates improvement.
Time Frame: Baseline to Week 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cutaneous flushing episodes
Arm/Group | Placebo Core Phase | Telotristat Etiprate 150 mg Core Phase | Telotristat Etiprate 250 mg Core Phase | Telotristat Etiprate 350 mg Core Phase | Telotristat Etiprate 500 mg Core Phase
Number analyzed (Participants) | 4 | 3 | 3 | 1 | 7
cutaneous flushing episodes | -0.43 (0.435) | -0.60 (1.044) | -0.30 (0.436) | -0.10 (0) | -0.03 (0.673)

7. Secondary Outcome: Change From Baseline in Severity of Abdominal Pain or Discomfort
Description: Participants recorded the severity of abdominal pain or discomfort in a daily diary assessed using a 4-point scale (0-none, 1-mild, 2-moderate, 3-severe). A negative change from Baseline indicates improvement.
Time Frame: Baseline to Week 4
Population: Participants from the mITT Set Core Phase, all participants who received any fraction of a dose of study drug and had at least 1 week of data recorded in the daily diary after receiving study drug, with data available for analysis. Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Core Phase | Telotristat Etiprate 150 mg Core Phase | Telotristat Etiprate 250 mg Core Phase | Telotristat Etiprate 350 mg Core Phase | Telotristat Etiprate 500 mg Core Phase
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 8
units on a scale | 0.04 (0.358) | 0.03 (0.586) | -0.53 (0.808) | 0.03 (0.153) | 0.16 (0.358)

8. Secondary Outcome: Change From Baseline in Urinary 5-hydroxyindoleacetic Acid (u5-HIAA)
Description: u5-HIAA is a standard test used in clinical practice to assess the neuroendocrine tumor (NET) activity and is collected as a 24-hour urine specimen. A negative change from Baseline indicates improvement.
Time Frame: Baseline to Week 4
Population: Participants from the Pharmacodynamic (PD) Analysis Set Core Phase, all participants who received any fraction of a dose of study drug and had a valid Baseline and at least 1 valid post-Baseline PD assessment, with data available for analysis.
Measure: Mean (Standard Deviation); unit: mg/24 hours
Arm/Group | Placebo Core Phase | Telotristat Etiprate 150 mg Core Phase | Telotristat Etiprate 250 mg Core Phase | Telotristat Etiprate 350 mg Core Phase | Telotristat Etiprate 500 mg Core Phase
Number analyzed (Participants) | 4 | 2 | 3 | 2 | 8
mg/24 hours | -20.73 (17.212) | -27.55 (45.891) | -0.67 (0.493) | 13.60 (19.092) | -35.49 (49.949)

9. Secondary Outcome: Change From Baseline in Chromogranin A
Description: Blood samples were collected for assessment of Chromogranin A level. A negative change from Baseline indicates improvement.
Time Frame: Baseline to Week 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Core Phase | Telotristat Etiprate 150 mg Core Phase | Telotristat Etiprate 250 mg Core Phase | Telotristat Etiprate 350 mg Core Phase | Telotristat Etiprate 500 mg Core Phase
Number analyzed (Participants) | 5 | 2 | 3 | 2 | 8
ng/mL | -3251.2 (7803.84) | -190.5 (225.57) | -12.3 (13.05) | 52.5 (60.10) | 26011.4 (59383.95)

10. Secondary Outcome: Number of Participants Reporting Improvement in the Subjective Global Assessment of Symptoms Associated With Carcinoid Syndrome
Description: Participants were asked to answer the following question: "In the past 7 days, have you had adequate relief of your carcinoid syndrome bowel complaints such as diarrhea, urgent need to have a bowel movement, abdominal pain, or discomfort?". The number of participants who answered Yes are reported.
Time Frame: Week 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Core Phase | Telotristat Etiprate 150 mg Core Phase | Telotristat Etiprate 250 mg Core Phase | Telotristat Etiprate 350 mg Core Phase | Telotristat Etiprate 500 mg Core Phase
Number analyzed (Participants) | 4 | 2 | 3 | 2 | 7
Participants | 0 | 1 | 2 | 1 | 3

11. Secondary Outcome: Change From Baseline in Frequency of Rescue for Short-acting Octreotide Use/Day
Description: Participants recorded details (location and frequency of injection) of subcutaneous injections of rescue, short-acting octreotide, if taken, in the daily diary. A negative change from Baseline indicates improvement.
Time Frame: Baseline to Week 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: injections per day
Arm/Group | Placebo Core Phase | Telotristat Etiprate 150 mg Core Phase | Telotristat Etiprate 250 mg Core Phase | Telotristat Etiprate 350 mg Core Phase | Telotristat Etiprate 500 mg Core Phase
Number analyzed (Participants) | 4 | 3 | 3 | 1 | 7
injections per day | -0.38 (0.695) | -0.03 (0.058) | 0.03 (0.058) | 0.00 (0) | -0.29 (0.669)

12. Secondary Outcome: Time to First Rescue, Short-acting Octreotide
Description: Time to the first subcutaneous injections of rescue, short-acting octreotide was determined from the participant's daily diary.
Time Frame: Baseline to Week 4
Population: Participants from the mITT Set Core Phase, all participants who received any fraction of a dose of study drug and had at least 1 week of data recorded in the daily diary after receiving study drug, As per protocol only the Placebo Core Phase and Telotristat Etiprate 500 mg Core Phase were included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo Core Phase | Telotristat Etiprate 500 mg Core Phase
Number analyzed (Participants) | 5 | 9
days | 1.00 [1.00 to NA] — The upper limit of 95% Confidence Interval was not obtained due to the low number of participants with events. | 1.00 [1.00 to NA] — The upper limit of 95% Confidence Interval was not obtained due to the low number of participants with events.

13. Secondary Outcome: Number of Participants Experiencing Complete Response at Week 4
Description: Complete Response to treatment was defined as one of the following: 1. Less than 4 bowel movements per day; or 2. A decrease in daily bowel movements that is ≥ 50% from baseline; or 3. A positive response to the global assessment question ("In the past 7 days, have you had adequate relief of your carcinoid syndrome bowel complaints such as diarrhea, urgent need to have a bowel movement, abdominal pain or discomfort?") for each of the last 2 weeks of the Treatment Period.
Time Frame: Baseline to Week 4
Population: The mITT Set Core Phase included all participants who received any fraction of a dose of study drug and had at least 1 week of data recorded in the daily diary after receiving study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Core Phase | Telotristat Etiprate 150 mg Core Phase | Telotristat Etiprate 250 mg Core Phase | Telotristat Etiprate 350 mg Core Phase | Telotristat Etiprate 500 mg Core Phase
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 9
Participants | 0 | 1 | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the core phase over 4 weeks and up to 180 weeks in the extension phase
Description: Safety Set included all participants who received at least one dose of study drug.
Arm/Group | Placebo Core Phase | Telotristat Etiprate 150 mg Core Phase | Telotristat Etiprate 250 mg Core Phase | Telotristat Etiprate 350 mg Core Phase | Telotristat Etiprate 500 mg Core Phase | Telotristat Etiprate Open-Label Extension Phase
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3 | 0/3 | 0/3 | 0/9 | 1/19
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3 | 0/3 | 1/3 | 0/9 | 8/19
Other Adverse Events (participants affected / at risk) | 4/5 | 3/3 | 3/3 | 2/3 | 9/9 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Core Phase (N=5) | Telotristat Etiprate 150 mg Core Phase (N=3) | Telotristat Etiprate 250 mg Core Phase (N=3) | Telotristat Etiprate 350 mg Core Phase (N=3) | Telotristat Etiprate 500 mg Core Phase (N=9) | Telotristat Etiprate Open-Label Extension Phase (N=19)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Mass excision (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal resection (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Core Phase (N=5) | Telotristat Etiprate 150 mg Core Phase (N=3) | Telotristat Etiprate 250 mg Core Phase (N=3) | Telotristat Etiprate 350 mg Core Phase (N=3) | Telotristat Etiprate 500 mg Core Phase (N=9) | Telotristat Etiprate Open-Label Extension Phase (N=19)
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 4 | 10
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 4 | 9
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 3
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 2
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 2 | 7
Early satiety (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 7
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 6
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 4
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 3
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 4
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 2
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 3
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Keratoconjunctivitis sicca (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Steatorrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Infusion site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vitamin A deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vitamin E deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal hypermotility (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phophatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Urine colour abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bilirubinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable subject matter.